CLINICAL TRIAL: NCT05264727
Title: Glucagon Suppression by Hyperglycemia in the Presence and Absence of Amino Acid Infusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22-000306; R01DK116231 (NIH)
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glucose; Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Adults, Obese Adults, Adults with Type 2 diabetes: Saline and Glucose (Experimental): Study visit: Subjects will receive a caffeine free, standardized evening meal and remain fasting overnight. An IV infusion of saline and glucose (50%) will be given the next morning and continue until the end of study. Blood draws will be collected frequently from the IV line to monitor blood glucose levels.
  Interventions: Drug: Dextrose
- Healthy Adults, Obese Adults, Adults with Type 2 diabetes: Amino Acid and Glucose (Experimental): Study visit: Subjects will receive a caffeine free, standardized evening meal and remain fasting overnight. An IV infusion of glucose (50%) will be given the next morning together with an IV infusion of Clinisol 15% (an amino acid mixture) will be given the next morning and continue until the end of study. Blood draws will be collected frequently from the IV line to monitor blood glucose levels.
  Interventions: Drug: Dextrose; Drug: Clinisol 15%

INTERVENTIONS:
Drug: Dextrose — Intravenous graded glucose infusion using 50% dextrose will commence at 1mg/kg/min and increase to 2 (0900), 4 (1000) and 8mg/kg/min (1100) every 60 minutes
Drug: Clinisol 15% — Intravenous infusion 0.003ml/kg/min infused from 0 to 240 minutes
  Other Names: Amino Acid Mixture
  Arms: Healthy Adults, Obese Adults, Adults with Type 2 diabetes: Amino Acid and Glucose

SUMMARY:
This study is being done to better understand how amino acids alter the release of glucagon and insulin compared to glucose alone in health and disease.

DETAILED DESCRIPTION:
T2DM and prediabetes are characterized by abnormal post-prandial suppression of glucagon, which contributes to postprandial hyperglycemia by increasing endogenous glucose production (EGP). In rodents, altered glucagon signaling changes α-cell function and mass - an effect mediated by changes in circulating AA concentrations. Are the elevated concentrations of branched-chain AA and other AA metabolites in T2DM a cause or an effect of global α-cell dysfunction? To measure glucagon secretion, as well as glucagon action, we have developed a population model of glucagon kinetics allowing us to deconvolve secretion from glucagon concentrations in a manner similar to Van Cauter's model for insulin secretion from C-peptide. This enables better characterization of α-cell function in humans. In addition to our novel methodology, we can characterize α-cell responsiveness to a graded glucose infusion, by quantifying (G50) - the change in glucose concentration necessary to suppress glucagon secretion by 50%. These experiments will determine if the glucagon secretion in response to AA differs in obese individuals with T2DM from that observed in obese individuals without T2DM.

ELIGIBILITY:
Inclusion Criteria - Obese Subjects with Type 2 Diabetes:

* HbA1c ≤ 8.5% (type 2 diabetic subjects).
* HbA1c ≤ 6.5% (obese and lean subjects).
* BMI ≥ 28 Kg/M^2 (Obese subjects with and without type 2 diabetes).
* BMI ≤ 25 Kg/M^2 (Lean subjects without type 2 diabetes).
* Use of sulfonylureas or metformin only (type 2 diabetec subjects).
* For female subjects: negative pregnancy test at the time of enrollment or study.
* No history of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* No active systemic illness or malignancy.
* No symptomatic macrovascular or microvascular disease.
* No contraindications to MRI (e.g., metal implants, claustrophobia).
* Hematocrit > 35%.
* TSH > 0.4 or < 5.5.
* Consumption of < 2 alcohol drinks per day or < 14 per week or a negative AUDIT questionnaire.

Exclusion Criteria - Obese Subjects with Type 2 Diabetes:

* HbA1c ³ 8.5%
* BMI ≤ 28 Kg/M2
* Use of insulin or agents other than sulfonylureas or metformin.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Contraindications to MRI (e.g., metal implants, claustrophobia).
* Hematocrit < 35%
* TSH < 0.4 or > 5.5.
* Consumption of > 2 alcohol drinks per day or > 14 per week or a positive AUDIT questionnaire.

Inclusion Criteria - Obese Subjects without Type 2 Diabetes:

* BMI ≥ 28 Kg/M2.
* > 5% liver fat content, as determined by MRI using the proton density fat fraction (PDFF) technique.

Exclusion Criteria - Obese Subjects without Type 2 Diabetes:

* HbA1c ≥ 6.5%
* BMI ≤ 28 Kg/M2
* Use of any glucose-lowering agents including metformin or sulfonylureas.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Contraindications to MRI (e.g., metal implants, claustrophobia).
* Hematocrit < 35%
* TSH < 0.4 or > 5.5.
* Consumption of > 2 alcohol drinks per day or > 14 per week or a positive AUDIT questionnaire.

Inclusion Criteria - Lean subjects without Diabetes:

- BMI ≤ 25 Kg/M^2).

Exclusion Criteria - Lean Subjects without Diabetes:

* HbA1c ≥ 6.5%.
* BMI ≥ 25 Kg/M^2.
* Use of any glucose-lowering agents including metformin or sulfonylureas.
* For female subjects: positive pregnancy test at the time of enrollment or study.
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Contraindications to MRI (e.g., metal implants, claustrophobia).
* Hematocrit < 35%.
* TSH < 0.4 or > 5.5.
* Consumption of > 2 alcohol drinks per day or > 14 per week or a positive AUDIT questionnaire.
* Liver fat content ≥ 5% as determined by MRI using the proton density fat fraction (PDFF) technique.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Glucagon Suppression (G50) caused by amino acids vs. saline | 240 minutes of study
  concentration of glucose necessary to suppress glucagon by 50%

SECONDARY OUTCOMES:
Glucagon suppression (G50) is greater in people with T2DM | 240 minutes of study
  concentration of glucose necessary to suppress glucagon by 50%
glucagon suppression (G50) is greater in obese compared to lean people without T2DM | 240 minutes of study
  concentration of glucose necessary to suppress glucagon by 50%

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials